CLINICAL TRIAL: NCT07210801
Title: Magnitude of Alignment With ESC Guidelines in Implantation Techniques of Cardiac Implantable Electronic Devices and Its Impact on Clinical Outcomes
Brief Title: CIED Implantation Technique at Assiut University Heart Hospital in Relation to ESC Guidelines
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Nagaty Ayoup Qods, Doctor, Assiut University
Other Study IDs: CIED Implantation Technique
Record Dates: First submitted 2025-09-18; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: CIED-related Infections; CIED Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CIEDimplantation — Compare current procedural CIED practice at AUHH to recent ESC guidelines.

SUMMARY:
This prospective observational cohort study will evaluate the extent to which cardiac implantable electronic device (CIED) implantation techniques at Assiut University Heart Hospital (AUHH) align with the evidence-based recommendations of the European Society of Cardiology (ESC).

DETAILED DESCRIPTION:
There is a huge and growing body of evidence demonstrating the importance of cardiac implantable electronic devices (CIEDs) in improving quality of life and survival among specific groups of patients with heart disease. This has led to an increasing number of implanted CIEDs, with approximately 1.2-1.4 million procedures performed annually worldwide. Over the years, advancements in device technology and implantation techniques have significantly improved patient outcomes and device longevity.

However, variations in implantation practices persist across different centers due to differences in training, available resources, and institutional protocols. The European Society of Cardiology (ESC) has established evidence-based guidelines outlining the optimal technique for CIED implantation, aiming to standardize practices and minimize procedure-related complications. These guidelines cover various aspects of the implantation process, including pre-procedural assessment, choice of venous access, lead positioning, infection prevention strategies, and post-implantation follow-up.

At Assiut University Heart Hospital, CIED implantation is routinely performed; however, the extent to which current practice aligns with the ESC-recommended optimal technique remains unclear. Understanding this alignment is crucial, as deviations from best practices may contribute to avoidable early complications, suboptimal device function, or reduced patient satisfaction.

This study aims to compare the current pacemaker implantation technique utilized at Assiut University Heart Hospital with the optimal implantation approach outlined in the latest ESC guidelines. Furthermore, it seeks to assess whether discrepancies or variations in CIED implantation techniques translate into differences in outcomes and complication rates. Assessing the degree of adherence to international guidelines by identifying gaps and areas for improvement may contribute to enhancing procedural quality, efficiency, patient safety, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All addult patients (≥18 years) referred foran indicatedCIED implantation at Assiut University Heart Hospital

Exclusion Criteria:

* Previous implantation of CIED implantation
* General contraindications of CIED
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will involve adult patients (≥18 years) receiving CIED for standard arrhythmic, conduction system diseases or heart failure indications over a period of two years,
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedure-related early complications (composite) | 30 day
  Percentage of patients who develop any of the following within 30 days after pacemaker implantation: hematoma requiring intervention, lead dislodgement requiring reintervention, pneumothorax requiring treatment, pocket or device-related infection requiring antibiotics or device removal, acute pacing failure or sensing abnormality requiring reintervention

SECONDARY OUTCOMES:
Incidence of late complications after pacemaker implantation | 12 month
  Number and percentage of patients who develop late device-related complications such as pocket erosion, late infection, venous thrombosis, or lead malfunction after 30 days and up to 12 months post-implantation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayes DL, Furman S. Cardiac pacing: how it started, where we are, where we are going. J Cardiovasc Electrophysiol. 2004 May;15(5):619-27. doi: 10.1046/j.1540-8167.2004.04088.x. No abstract available. PMID 15149441
- [Result] Da Costa A, Kirkorian G, Isaaz K, Touboul P. [Secondary infections after pacemaker implantation]. Rev Med Interne. 2000 Mar;21(3):256-65. doi: 10.1016/s0248-8663(00)80045-4. French. PMID 10763187
- [Result] Kranick S, Mishra N, Theertham A, Vo H, Hiltner E, Coromilas J, Kassotis J. A Survey of Antibiotic Use During Insertion of Cardiovascular Implantable Devices Among United States Implanters. Angiology. 2023 Apr;74(4):351-356. doi: 10.1177/00033197221114689. Epub 2022 Jul 11. PMID 35816293